CLINICAL TRIAL: NCT05816499
Title: A Phase Ib/II Trial of Cadonilimab (PD-1/CTLA-4 Bispecific Antibody) in Combination With Anlotinib and Docetaxel in Patients (Pts) With Checkpoint Inhibitor (CPI)-Experienced Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: Cadonilimab in Patients (Pts) With Advanced Non-small Cell Lung Cancer (NSCLC)
Acronym: AK104IIT018
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: The Affiliated Hospital of Qingdao University (Other); Anhui Provincial Hospital (Other Government); Zhejiang University (Other)
Responsible Party: Principal Investigator, Baohui Han, chief physician, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-018
Record Dates: First submitted 2023-03-01; First posted 2023-04-18 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: NSCLC Stage IV; NSCLC Stage IIIB; NSCLC Stage IIIC
Keywords: Cadonilimab; AK104; NSCLC; resistance
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anlotinib; Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm A (cadonilimab，anlotinib，docetaxel ) (Experimental): Patients receive anlotinib 6mg/8mg/10mg qd 2W/3W and cadonilimab IV over 90 minutes on day 1. Patients also receive docetaxel 60-75 mg/m2 IV over 60 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cadonilimab; Drug: Anlotinib; Drug: Docetaxel

INTERVENTIONS:
Drug: Cadonilimab — Given IV, 10mg/kg Q3W
  Other Names: AK104
Drug: Anlotinib — oral，6mg/8mg/10mg qd 2W/3W
  Other Names: AL3818
Drug: Docetaxel — Given IV, 60-75mg/m2 Q3W
  Other Names: Docetaxel Trihydrate; Docetaxel Hydrate; Taxoltere Metro; RP 56976; RP-56976; RP56976; Docetaxel Anhydrous; N-Debenzoyl-N-tert-butoxycarbonyl-10-deacetyltaxol; N Debenzoyl N tert butoxycarbonyl 10 deacetyltaxol; NSC 628503; Taxotere

SUMMARY:
This phase Ib/II trial studies how well cadonilimab combined with anlotinib and docetaxel work in treating patients with non-small cell lung cancer that is stage IV or has come back. Cadonilimab, a PD-1/CTLA-4 bispecific antibody, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Anlotinib can regulate tumor microenvironment. Docetaxel was used in standard of care chemotherapy for non-small cell lung cancer, work to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving cadonilimab, anlotinib and docetaxel together may work better in treating patients with non-small lung cancer compared to standard of care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. Dose discovery stage: evaluate the safety of cadonilimab combined with anlotinib and docetaxel in the treatment of locally advanced and metastatic NSCLC after failure of treatment with PD-L1/1 inhibitors and the recommended dose of anlotinib.
2. Dose expansion stage: evaluate the 6-month PFS rate of patients with locally advanced and metastatic NSCLC after failure of treatment with PD-L1/1 inhibitors by cadonilimab combined with anlotinib and docetaxel, which was evaluated by researchers based on RECIST v1.1.

SECONDARY OBJECTIVES:

1. evaluate the objective response rate (ORR), progression-free survival (PFS), disease control rate (DCR), duration of response (DoR), time to response (TTR), and total survival (OS) of patients with locally advanced and metastatic NSCLC after failure of treatment with PD-L1/1 inhibitors with cadonilimab, anlotinib, and docetaxel.
2. evaluate the safety and tolerability of cadonilimab combined with arotinib and docetaxel in the treatment of locally advanced and metastatic NSCLC after failure of treatment with PD-L1/1 inhibitor.

OUTLINE:

This is a prospective, open, single-arm, multi-center, phase I b/II clinical study. All patients were confirmed Locally advanced (stage IIIB/IIIC) that cannot be resected by radical surgery and cannot accept radical synchronous/sequential radiotherapy and chemotherapy or metastatic (stage IV) NSCLC by histology or cytology. Patients must have progressed on at most a PD-1/L1 inhibitor and a platinum-based chemotherapy (combined or sequential, regardless of sequence), and at least two cycles of PD-1/L1 inhibitor (combined or non-combined chemotherapy) with clinical benefits (PFS ≥ 3 months). The study is divided into two parts. The first part is the dose discovery stage. The patients will receive a 21-day observation period of dose limiting toxicity (DLT). 3-6 subjects will be enrolled in each dose, and finally evaluate the safety and determine the recommended dose (RP2D) for phase II clinical study according to the "3+3" principle. We will continue to recruit 44 patients at the dose expansion stage.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years old
2. Locally advanced (stage IIIB/IIIC) that cannot be resected by radical surgery and cannot accept radical synchronous/sequential radiotherapy and chemotherapy and metastatic (stage IV) NSCLC confirmed by histology or cytology
3. Patients must have progressed on at most a PD-1/L1 inhibitor and a platinum-based chemotherapy (combined or sequential, regardless of sequence), and at least two cycles of PD-1/L1 inhibitor (combined or non-combined chemotherapy) with clinical benefits (PFS ≥ 3 months)
4. Patients must not have EGFR sensitizing mutations, EGFR T790M mutation, ALK gene fusion, and ROS 1 gene rearrangement, and BRAF V600E mutation.
5. Has measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
6. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
7. Life expectancy > 12 weeks as determined by the investigator
8. Patients must have at least one measurable lesion (as defined by RECIST v1.1), which is suitable for repeated and accurate measurement
9. Absolute neutrophil count (ANC) ≥ 1500/uL (collected within 10 days prior to the start of study treatment)
10. Platelets ≥ 100 000/uL (collected within 10 days prior to the start of study treatment)
11. Hemoglobin ≥ 9.0 g/dL (collected within 10 days prior to the start of study treatment)
12. Creatinine clearance [CrCl]) ≥ 50 mL/min(Creatinine clearance (CrCl) should be calculated per institutional standard)
13. Total bilirubin ≤ 1.5 x ULN (collected within 10 days prior to the start of study treatment)
14. Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 2.5 x ULN (≤ 5 x ULN for participants with liver metastases) (collected within 10 days prior to the start of study treatment
15. Serum albumin(ALB)≥28 g/L
16. International standardized ratio (INR) and activated partial thrombin time (APTT) ≤ 1.5 × ULN
17. Left ventricular ejection fraction (LVEF) ≥ 50%
18. A male participant must agree to use a contraception during the treatment period plus an additional 120 days after the last dose of study treatment and refrain from donating sperm during this period
19. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    1. Not a woman of childbearing potential (WOCBP) OR
    2. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days plus 30 days (a menstruation cycle) after the last dose of study treatment

Exclusion Criteria:

1. Previously received treatment for tumor immune mechanism other than any anti-PD-1/L1 inhibitor for advanced NSCLC stage, such as CTLA-4（CD152）、TIGIT、OX-40、CD137、ICOS、CD40、CD47、CD73、GITR、TOX、LAG-3、TIM3、SIRPα、BTLA（CD272）、VISTA（B7-H5）、LIGHT（CD258）、B7-H3（CD276）、 B7-H4（VTCN1）、HVEM、CD80/CD86、MHC Ⅱ、GAL9、IDO、PVR（CD155）、Nectin-2（CD112）.
2. Patients have prior exposure to docetaxel, anlotinib, lenvatinib, apatinib, cabozantinib.
3. The last systemic anti-tumor treatment (chemotherapy, immunotherapy, biological agents, anti-angiogenic drugs, etc.) was received within 3 weeks before the first administration.
4. The following treatments were received within 2 weeks before the first administration: TKI treatment, hormone anti-tumor treatment, palliative local treatment for non-target lesions Non-specific immunomodulatory therapy (such as interleukin, interferon, thymosin, tumor necrosis factor, etc., excluding IL-11 for thrombocytopenia).
5. Patients with explosive progress.
6. Patients with other active malignant tumors except for NSCLC within 3 years before enrollment. Patients with other malignant tumors that have been cured by local treatment, such as basal or cutaneous squamous cell carcinoma, superficial bladder cancer cancer, cervical or breast cancer in situ, are not excluded.
7. Patients with active autoimmune diseases that require systemic treatment in the past two years (such as the use of disease improvement drugs, corticosteroids, immunosuppressants) (excluding irAE caused by the use of PD-1/L1 inhibitors). Replacement therapy (such as thyroid hormone, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered as a systemic treatment.
8. Patients can not swallow pills, with malabsorption syndrome, or any condition that affects gastrointestinal absorption;
9. Patients with active or previous history of inflammatory bowel disease (such as Crohn's disease, ulcerative colitis or chronic diarrhea).
10. Patients have a history of immune deficiency, with HIV antibody test positive or use systemic corticosteroids or other immunosuppressants for a long time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
RP2D of anlotinib | Up to 21 days after the first cycle of study treatment
  Will be evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Overall toxicity incidence as well as toxicity profiles will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses. Proportion of acute and late toxicity will be reported, and 95% confidence intervals will be estimated using the Clopper-Pearson method.
6-month progression-free survival (PFS) rate | up to 6 months
  Will be determined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Will be reported and its 95% confidence intervals will be estimated using the Clopper-Pearson method. PFS rates of two patient groups stratified by binary biomarker (PD-L1 and KRAS status), respectively will be estimated with the Kaplan-Meier method and compared using the log-rank test, respectively. Cox proportional hazards models will be further used in the multivariable analyses to assess adjusted effect of PD-L1 and KRAS status on the patients' PFS after adjusting for other factors. Interaction terms between these factors will also be tested for statistical significance. The proportional hazards assumption will be evaluated graphically and analytically with regression diagnostics. Violations of the proportional hazards assumptions will be addressed by use of time-dependent covariates or extended Cox regression models.

SECONDARY OUTCOMES:
Overall response rate | Through study completion, an average of 1 year
  Will be determined per RECIST 1.1 and immune-modified Response Evaluation Criteria in Solid Tumors.
Overall survival (OS) | up to 10 years
  OS and rates of two patient groups stratified by binary biomarker (PD-L1 and KRAS status), respectively will be estimated with the Kaplan-Meier method and compared using the log-rank test, respectively. Cox proportional hazards models will be further used in the multivariable analyses to assess adjusted effect of PD-L1 and KRAS status on the patients' OS after adjusting for other factors. Interaction terms between these factors will also be tested for statistical significance. The proportional hazards assumption will be evaluated graphically and analytically with regression diagnostics. Violations of the proportional hazards assumptions will be addressed by use of time-dependent covariates or extended Cox regression models.
Investigator assessed-progression-free survival (IA-PFS) | From date of sub-study registration to date of first documentation of progression assessed by central review or symptomatic deterioration, or death due to any cause, assessed up to 3 years
  Will be estimated using the method of Kaplan-Meier. Median and landmark time-point estimates will be based on the Kaplan-Meier estimates. The average hazard ratio (HR) will be estimated using a Cox proportional hazards model. An assessment of the proportional hazards assumption will be performed and an assessment of the time-dependent HR will be done.
Incidence of adverse events | Up to 30 days after the last dose of study treatment
  Will be evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Overall toxicity incidence as well as toxicity profiles will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses. Proportion of acute and late toxicity will be reported, and 95% confidence intervals will be estimated using the Clopper-Pearson method.

CONTACTS AND LOCATIONS:
Overall Officials: Baohui Han, M.D, Study Chair — ShanghaiChest Hospital; Jianya Zhou, M.D, Principal Investigator — Zhejiang University; Zhuang Yu, M.D, Principal Investigator — The Affiliated Hospital of Qingdao University; Jing Wang, M.D, Principal Investigator — The Affiliated Hospital of Qingdao University; lejie Cao, M.D, Principal Investigator — Anhui Provincial Hospital
Locations (5):
- China (5):
  - lejie Cao, Hefei, Anhui
  - Jing Wang, Qingdao, Shandong
  - Zhuang Yu, Qingdao, Shandong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Jianya Zhou, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication

REFERENCES:
- [Background] Travis WD, Brambilla E, Noguchi M, Nicholson AG, Geisinger KR, Yatabe Y, Beer DG, Powell CA, Riely GJ, Van Schil PE, Garg K, Austin JH, Asamura H, Rusch VW, Hirsch FR, Scagliotti G, Mitsudomi T, Huber RM, Ishikawa Y, Jett J, Sanchez-Cespedes M, Sculier JP, Takahashi T, Tsuboi M, Vansteenkiste J, Wistuba I, Yang PC, Aberle D, Brambilla C, Flieder D, Franklin W, Gazdar A, Gould M, Hasleton P, Henderson D, Johnson B, Johnson D, Kerr K, Kuriyama K, Lee JS, Miller VA, Petersen I, Roggli V, Rosell R, Saijo N, Thunnissen E, Tsao M, Yankelewitz D. International association for the study of lung cancer/american thoracic society/european respiratory society international multidisciplinary classification of lung adenocarcinoma. J Thorac Oncol. 2011 Feb;6(2):244-85. doi: 10.1097/JTO.0b013e318206a221. PMID 21252716
- See also: 2021 ESMO Abstract #1191O — https://www.esmo.org/
- See also: 2021 ESMO Abstract #1284P — https://www.esmo.org/